CLINICAL TRIAL: NCT04819022
Title: Digitally Assisted Rehabilitation Programs for Musculoskeletal Disorders: a Large-scale, Multi-disorder, Prospective, Longitudinal Cohort Study
Brief Title: SWORD Health Patient Registry
Status: Completed | Type: Observational
Sponsor: Sword Health, SA (Industry)
Responsible Party: Sponsor
Other Study IDs: SH-MSD-OBS-01
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Musculoskeletal Diseases
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Subacute Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Musculoskeletal disorder
  Interventions: Device: Acute and post-acute; Device: Chronic; Device: Post-surgical

INTERVENTIONS:
Device: Acute and post-acute — These programs will cover patients suffering from acute or post-acute musculoskeletal conditions including, but not limited to, shoulder pain (tendinitis/impingement/bursitis), neck pain, low back pain, knee or hip pain/osteoarthritis, which significantly impact their quality of life, to the extent they seek specialised care in direct relation to these disorders.
Device: Chronic — These programs will cover patients suffering from chronic musculoskeletal conditions including, but not limited to, shoulder pain (tendinitis/impingement/bursitis), neck pain, low back pain, knee or hip pain/osteoarthritis, which significantly impact their quality of life, to the extent they seek specialised care in direct relation to these disorders.
Device: Post-surgical — These programs will cover patients submitted to surgery for a given musculoskeletal condition, including, but not limited to, shoulder tendon repair, shoulder replacement, spinal surgery, hip or knee replacement, meniscal repair, knee ligament reconstruction, undergoing physical rehabilitation programs after surgery.

SUMMARY:
The purpose of this study is to create a research repository, comprised of data collected in the course of physical rehabilitation programs for musculoskeletal disorders (MSDs) using the medical device SWORD Phoenix®.

This will allow the company to ascertain the acceptance, engagement and effectiveness of programs using this asynchronous tele-rehabilitation platform in the treatment of multiple MSDs.

DETAILED DESCRIPTION:
The data that will be collected in the scope of this registry includes:

1. data that is sourced from the subject, which will be collected by the physical therapist managing that subject;
2. data that is generated by the physical therapist through interaction with the web-based Portal (i.e. session composition in terms of exercises, sets, repetitions, usage or not of external resistance)
3. data that is generated by the subject through interaction with the app (i.e. pain and fatigue levels, satisfaction)
4. data that is generated automatically by the medical device (i.e. range of motion, compliance)

Collection and objective analysis of the collected data will allow:

1. Assess the adoption, engagement and feasibility of digital care programs for musculoskeletal conditions and musculoskeletal health
2. Assess the results of digital care programs and compare the costs with the benefits obtained;
3. Correlate the results with patient's demographic and clinical profiles;
4. Examine the impact of mental health and the behavioral modification components of SWORD Health interventions on disease markers, comorbidities, and productivity;
5. Increase the knowledge on several musculoskeletal conditions, namely how they progress and respond to digital care programs;
6. Develop new or improved tools to assist clinicians in the management of these conditions and in helping people achieve better musculoskeletal health

Clinical outcomes

The primary outcome will be the evolution of patient's clinical condition along the rehabilitation program, objectively estimated through the monitoring data collected using SWORD Phoenix®, as part of patients' supervision routine. Depending on the condition, primary and secondary outcome measures vary.

In any case, this registry will include a complete characterisation of the clinical condition, as well as the periodic assessment of: a) joints' range of motion (collect by the medical device); b) performance indicators (through condition-specific tests); c) patient-reported outcomes (obtained using internationally validated pathology-specific questionnaires); d) pain and fatigue levels (reported by patients by the end of each therapeutic exercise session); e) compliance; f) patient satisfaction

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old;
* Initiating a rehabilitation program using the medical device SWORD Phoenix®;
* Able to understand study procedures and willing to provide informed consent.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: These programs will cover patients suffering from musculoskeletal conditions including, but not limited to, shoulder pain (tendinitis/impingement/bursitis), neck pain, low back pain, knee or hip pain/osteoarthritis, which, irrespective of their duration (acute, post-acute or chronic), significantly impact their quality of life, to the extent they seek specialized care in direct relation to these disorders. The programs will also cover patients submitted to surgery for a given musculoskeletal condition, including, but not limited to, shoulder tendon repair, shoulder replacement, spinal surgery, hip or knee replacement, meniscal repair, knee ligament reconstruction, undergoing physical rehabilitation programs after surgery.
Sampling Method: Probability Sample
Enrollment: 10500 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Timed-up-and-go test (TUG) | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change in condition-specific clinical outcomes over time measured through the TUG test. The TUG consists on the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. As a reference, patients treated with conventional physiotherapy 6 months after total knee replacement reported a TUG of 9.1 seconds.
Foot and Ankle Ability Measure (FAAM) | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change in condition-specific clinical outcomes over time, measured through the Foot and Ankle Ability Measure (FAAM).
  FAAM is a self-report measure that assesses physical function of individuals with lower leg, foot, and ankle musculoskeletal disorders. Thus instrument included 2 subscales: 1) Activities of Daily Living (ADLs) with 21 items and 2) Sports with 8 items. For each subscale patients are asked to answer each question with a single response that most clearly describes their condition within past week. To calculate the score for either subscale, the total number of points are added, divided by the total number os possible points (ADLs-84; Sports-32) and then multiplied by 100.
Constant-Murley Shoulder Outcome Score (CM) | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change in condition-specific clinical outcomes over time, measured through the CM score.
  The scale consists of:
  1. Subjective variables: a) Pain - Absence of pain gets maximum score of 15; b) Limitation of Activities of daily living (sleep, work, recreation/sport). No limitations get maximum score, 20. The subjective variables add to a maximum score of 35.
  2. Objective variables: c) Range of motion - Maximum score 40; d) Strength - Maximum Score 25 Objective variables add to a total of 65. Total Constant Score is calculated by adding the scores from subjective and objective variables. The maximum possible total score is 100.
Oswestry Disability Index (ODI) | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change in condition-specific clinical outcomes over time measured through the Oswestry Disability Index (ODI). \ The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.
Knee range of motion | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change in meniscal repair or cruciate ligament reconstruction patients' clinical outcomes over time measured through knee range of motion (ROM) (flexion/extension/abduction/rotation), in degrees, as directly retrieved from the angle measurement tool integrated within the medical device.

SECONDARY OUTCOMES:
Neck, lower spine, shoulder, elbow, ankle, hip and knee range of motion (ROM) | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change in condition-specific clinical outcomes over time measured through Neck, lower spine, shoulder, elbow, ankle, hip and knee range of motion (ROM) (flexion/extension/abduction/rotation), in degrees, as directly retrieved from the angle measurement tool integrated within the medical device.
Short version of the Disabilities of the Arm, Shoulder and Hand questionnaire | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change in condition-specific clinical outcomes over time measured through the short version of the Disabilities of the Arm, Shoulder and Hand questionnaire (QuickDASH).
  Scoring Formula = ([(sum of n responses)/n] -1)x(25).
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change in condition-specific clinical outcomes over time measured through the Knee Injury and Osteoarthritis Outcome Score (KOOS) Scoring Formula: 100 - [(patient's score of the subscale x 100)/(total score of the subscale)]
Hip Disability and Osteoarthritis Outcome Score | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change in condition-specific clinical outcomes over time measured through the hip disability and osteoarthritis outcome score (HOOS) Scoring Formula: 100 - [(patient's score of the subscale x 100)/(total score of the subscale)]
Fear avoidance behaviour | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change over time in clinical outcomes common to all conditions measured through the Fear Avoidance Beliefs Questionnaire - Work & Physical Activity (FABQ).
Single leg stance test (SLS) | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change in condition-specific clinical outcomes over time measured through the SLS test. Used to assess static postural and balance control. Performed with eyes open and hands on the hips. Patient must stand unassisted on one leg, timed from the time the other foot leaves the ground till when the foot touches the ground again or the arms leave the hips. If unable to stand for 5 seconds or less client at greater risk of injury from fall.
Self-reported Pain (NPRS) | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change over time in clinical outcomes common to all conditions measured through a 0-10 Pain Numerical Rating Scale
Self-reported Pain (VAS) | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change over time in clinical outcomes common to all conditions measured through a 0-10 Visual Analogue Scale for pain
Self-reported fatigue (VAS) | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change over time in clinical outcomes common to all conditions measured through a 0-10 Visual Analogue Scale for fatigue
Self-reported satisfaction | Each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Self-reported at the end of the program through the question: "On a scale from 0 to 10, how likely is it that you would recommend this intervention to a friend or neighbour?"
Compliance | Each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Average number os sessions performed per week

CONTACTS AND LOCATIONS:
Overall Officials: Fernando D Correia, MD, Principal Investigator — SWORD Health, Inc
Locations (1):
- SWORD Health, S.A., Porto, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and study aggregate results (including anonymised individual patient data) will be made available.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available upon studies publication, for 5 years.
Access Criteria: Study protocol will be available through a direct link in this platform. The excel file with the aggregate results will be made available as supplementary information upon study publication

REFERENCES:
- [Derived] Correia FD, Molinos M, Neves C, Janela D, Carvalho D, Luis S, Francisco GE, Lains J, Bento V. Digital Rehabilitation for Acute Ankle Sprains: Prospective Longitudinal Cohort Study. JMIR Rehabil Assist Technol. 2021 Sep 30;8(3):e31247. doi: 10.2196/31247. PMID 34499038